CLINICAL TRIAL: NCT01516879
Title: A Double-Blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate Long-Term Tolerability and Durable Efficacy of AMG 145 (Evolocumab) on LDL-C in Hyperlipidemic Subjects
Brief Title: Durable Effect of PCSK9 Antibody CompARed wiTh placEbo Study
Acronym: DESCARTES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110109
Record Dates: First submitted 2012-01-18; First posted 2012-01-25 (Estimated); Results first posted 2015-09-29 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Hypercholesterolemia
Keywords: Cholesterol; High Cholesterol; Elevated Cholesterol; Raised Cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — evolocumab; Atorvastatin; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Evolocumab (Experimental): Participants received evolocumab 420 mg subcutaneously once a month for 52 weeks in addition to background lipid-lowering therapy.
  Interventions: Biological: Evolocumab; Drug: Atorvastatin; Drug: Ezetimibe; Other: Diet Only
- Placebo (Placebo Comparator): Participants received placebo subcutaneously once a month for 52 weeks in addition to background lipid-lowering therapy.
  Interventions: Biological: Placebo; Drug: Atorvastatin; Drug: Ezetimibe; Other: Diet Only

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection once a month
  Other Names: AMG 145; Repatha
  Arms: Evolocumab
Biological: Placebo — Administered by subcutaneous injection once a month
  Arms: Placebo
Drug: Atorvastatin — Background lipid lowering therapy: 10 mg or 80 mg atorvastatin orally once daily.
Drug: Ezetimibe — Background lipid lowering therapy: ezetimibe 10 mg orally once a day
Other: Diet Only — Diet only, no lipid lowering background drug given

SUMMARY:
To evaluate the efficacy, safety, and tolerability of 52 weeks of subcutaneous (SC) evolocumab (AMG 145) compared with placebo when added to assigned background lipid-lowering therapy.

DETAILED DESCRIPTION:
Eligible participants with screening central laboratory low-density lipoprotein cholesterol (LDL-C) values ≥ 75 mg/dL (1.9 mmol/L) were instructed to follow National Cholesterol Education Program (NCEP) Adult Treatment Panel III (ATP) Therapeutic Lifestyle Changes (TLC) diet and were assigned to 1 of the following 4 background lipid-lowering therapies for a 4-week stabilization period based upon their screening LDL-C and its distance from the individual's required goal as stipulated by their NCEP ATP III risk category:

1. no drug therapy required - diet alone
2. low dose drug therapy required - diet plus atorvastatin 10 mg orally (PO) once daily (QD)
3. high dose drug therapy required - diet plus atorvastatin 80 mg PO QD
4. maximal drug therapy required - diet plus atorvastatin 80 mg PO QD plus ezetimibe 10 mg PO QD.

If the participant met entry criteria at the end of the lipid stabilization period they were randomized 2:1 to receive evolocumab 420 mg or placebo subcutaneously once a month for 52 weeks in addition to their background therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent.
* Fasting LDL-C ≥ 75 mg/dL and meeting the following LDL-C values on background lipid-lowering therapy:

  * < 100 mg/dL for subjects with diagnosed coronary heart disease (CHD) or CHD risk equivalent
  * < 130 mg/dL for subjects without diagnosed CHD or CHD risk equivalent
  * OR on maximal background lipid-lowering therapy defined as atorvastatin 80 mg PO QD and ezetimibe 10 mg PO QD
* Fasting triglycerides ≤ 400 mg/dL

Exclusion Criteria:

* New York Heart Association (NYHA) II-IV heart failure, or last known left ventricular ejection fraction < 30%
* Uncontrolled cardiac arrhythmia
* Myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or stroke within 3 months prior to randomization, type 1 diabetes, newly diagnosed or poorly controlled type 2 diabetes
* Uncontrolled hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 905 (Actual)
Dates: Start 2012-01-05 (Actual); Primary Completion 2013-10-14 (Actual); Study Completion 2013-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (85):
- United States (36):
  - Research Site, Birmingham, Alabama
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Encinitas, California
  - Research Site, Spring Valley, California
  - Research Site, Westlake Village, California
  - Research Site, DeLand, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Ponte Vedra, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Auburn, Maine
  - Research Site, Bethesda, Maryland
  - Research Site, Chevy Chase, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Brockton, Massachusetts
  - Research Site, Saint Paul, Minnesota
  - Research Site, Olive Branch, Mississippi
  - Research Site, Las Vegas, Nevada
  - Research Site, Endwell, New York
  - Research Site, New Windsor, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Renton, Washington
  - Research Site, Seattle, Washington
- Australia (6):
  - Research Site, Camperdown, New South Wales
  - Research Site, Maroubra, New South Wales
  - Research Site, Carina Heights, Queensland
  - Research Site, Milton, Queensland
  - Research Site, Fitzroy, Victoria
  - Research Site, Perth, Western Australia
- Austria (4):
  - Research Site, Feldkirch
  - Research Site, Innsbruck
  - Research Site, Salzburg
  - Research Site, Wels
- Belgium (6):
  - Research Site, AnthÃ©e
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Gozée
  - Research Site, Ham
  - Research Site, Ostend
- Canada (9):
  - Research Site, Victoria, British Columbia
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, Cambridge, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
- Czechia (7):
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, Hradec Králové
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Slaný
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Ballerup Municipality
  - Research Site, Vejle
- Hungary (6):
  - Research Site, Baja
  - Research Site, Budapest
  - Research Site, Komárom
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Zalaegerszeg
- South Africa (8):
  - Research Site, Lyttelton, Gauteng
  - Research Site, Chatsworth, Durban, KwaZulu-Natal
  - Research Site, eManzimtoti, KwaZulu-Natal
  - Research Site, Observatory, Western Cape
  - Research Site, Paarl, Western Cape
  - Research Site, Parow, Western Cape
  - Research Site, Somerset West, Western Cape
  - Research Site, Bloemfontein

REFERENCES:
- [Background] Toth PP, Sattar N, Blom DJ, Martin SS, Jones SR, Monsalvo ML, Elliott M, Davis M, Somaratne R, Preiss D. Effect of Evolocumab on Lipoprotein Particles. Am J Cardiol. 2018 Feb 1;121(3):308-314. doi: 10.1016/j.amjcard.2017.10.028. Epub 2017 Nov 8. PMID 29221604
- [Background] Blom DJ, Koren MJ, Roth E, Monsalvo ML, Djedjos CS, Nelson P, Elliott M, Wasserman SM, Ballantyne CM, Holman RR. Evaluation of the efficacy, safety and glycaemic effects of evolocumab (AMG 145) in hypercholesterolaemic patients stratified by glycaemic status and metabolic syndrome. Diabetes Obes Metab. 2017 Jan;19(1):98-107. doi: 10.1111/dom.12788. Epub 2016 Oct 14. PMID 27619750
- [Background] Blom DJ, Djedjos CS, Monsalvo ML, Bridges I, Wasserman SM, Scott R, Roth E. Effects of Evolocumab on Vitamin E and Steroid Hormone Levels: Results From the 52-Week, Phase 3, Double-Blind, Randomized, Placebo-Controlled DESCARTES Study. Circ Res. 2015 Sep 25;117(8):731-41. doi: 10.1161/CIRCRESAHA.115.307071. Epub 2015 Jul 30. PMID 26228031
- [Background] Blom DJ, Hala T, Bolognese M, Lillestol MJ, Toth PD, Burgess L, Ceska R, Roth E, Koren MJ, Ballantyne CM, Monsalvo ML, Tsirtsonis K, Kim JB, Scott R, Wasserman SM, Stein EA; DESCARTES Investigators. A 52-week placebo-controlled trial of evolocumab in hyperlipidemia. N Engl J Med. 2014 May 8;370(19):1809-19. doi: 10.1056/NEJMoa1316222. Epub 2014 Mar 29. PMID 24678979
- [Background] Daviglus ML, Ferdinand KC, Lopez JAG, Wu Y, Monsalvo ML, Rodriguez CJ. Effects of Evolocumab on Low-Density Lipoprotein Cholesterol, Non-High Density Lipoprotein Cholesterol, Apolipoprotein B, and Lipoprotein(a) by Race and Ethnicity: A Meta-Analysis of Individual Participant Data From Double-Blind and Open-Label Extension Studies. J Am Heart Assoc. 2021 Jan 5;10(1):e016839. doi: 10.1161/JAHA.120.016839. Epub 2020 Dec 16. PMID 33325247
- [Background] Kuchimanchi M, Grover A, Emery MG, Somaratne R, Wasserman SM, Gibbs JP, Doshi S. Population pharmacokinetics and exposure-response modeling and simulation for evolocumab in healthy volunteers and patients with hypercholesterolemia. J Pharmacokinet Pharmacodyn. 2018 Jun;45(3):505-522. doi: 10.1007/s10928-018-9592-y. Epub 2018 May 7. PMID 29736889
- [Background] Kasichayanula S, Grover A, Emery MG, Gibbs MA, Somaratne R, Wasserman SM, Gibbs JP. Clinical Pharmacokinetics and Pharmacodynamics of Evolocumab, a PCSK9 Inhibitor. Clin Pharmacokinet. 2018 Jul;57(7):769-779. doi: 10.1007/s40262-017-0620-7. PMID 29353350
- [Background] Sattar N, Toth PP, Blom DJ, Koren MJ, Soran H, Uhart M, Elliott M, Cyrille M, Somaratne R, Preiss D. Effect of the Proprotein Convertase Subtilisin/Kexin Type 9 Inhibitor Evolocumab on Glycemia, Body Weight, and New-Onset Diabetes Mellitus. Am J Cardiol. 2017 Nov 1;120(9):1521-1527. doi: 10.1016/j.amjcard.2017.07.047. Epub 2017 Jul 31. PMID 28844508
- [Background] Toth PP, Descamps O, Genest J, Sattar N, Preiss D, Dent R, Djedjos C, Wu Y, Geller M, Uhart M, Somaratne R, Wasserman SM; PROFICIO Investigators. Pooled Safety Analysis of Evolocumab in Over 6000 Patients From Double-Blind and Open-Label Extension Studies. Circulation. 2017 May 9;135(19):1819-1831. doi: 10.1161/CIRCULATIONAHA.116.025233. Epub 2017 Mar 1. PMID 28249876
- [Background] Toth PP, Jones SR, Monsalvo ML, Elliott-Davey M, Lopez JAG, Banach M. Effect of Evolocumab on Non-High-Density Lipoprotein Cholesterol, Apolipoprotein B, and Lipoprotein(a): A Pooled Analysis of Phase 2 and Phase 3 Studies. J Am Heart Assoc. 2020 Mar 3;9(5):e014129. doi: 10.1161/JAHA.119.014129. Epub 2020 Mar 2. PMID 32114889
- [Background] Wasserman SM, Sabatine MS, Koren MJ, Giugliano RP, Legg JC, Emery MG, Doshi S, Liu T, Somaratne R, Gibbs JP. Comparison of LDL-C Reduction Using Different Evolocumab Doses and Intervals: Biological Insights and Treatment Implications. J Cardiovasc Pharmacol Ther. 2018 Sep;23(5):423-432. doi: 10.1177/1074248418774043. Epub 2018 May 16. PMID 29768954
- [Background] Schludi B, Giugliano RP, Sabatine MS, Raal FJ, Teramoto T, Koren MJ, Stein EA, Wang H, Monsalvo ML. Time-averaged low-density lipoprotein cholesterol lowering with evolocumab: Pooled analysis of phase 2 trials. J Clin Lipidol. 2022 Jul-Aug;16(4):538-543. doi: 10.1016/j.jacl.2022.05.069. Epub 2022 Jun 6. PMID 35760720
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with fasting low-density lipoprotein cholesterol (LDL-C) ≥ 75 mg/dL and triglycerides ≤ 400 mg/dL were eligible. The first patient enrolled on 5 January 2012 and the last patient enrolled on 12 October 2012. All patients were counseled on the National Cholesterol Education Program Adult Treatment Panel III Therapeutic Lifestyle Changes diet.
Pre-assignment Details: Patients were assigned to 1 of 4 background lipid-lowering regimens for a 4-12 week stabilization period: diet alone, diet and 10 mg atorvastatin daily, diet and 80 mg atorvastatin daily, or diet, 80 mg atorvastatin and 10 mg ezetimibe daily. Patients meeting criteria were randomized 2:1 to evolocumab or placebo, stratified by background therapy.
Period: Overall Study
Arm/Group | Placebo | Evolocumab
Started | 303 | 602
Received Treatment | 302 | 599
Completed | 287 | 568
Not Completed | 16 | 34
Not completed — Withdrawal by Subject | 9 | 11
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 2 | 11
Not completed — Other | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Evolocumab | Total
Number analyzed (Participants) | 303 | 602 | 905
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (10.3) | 55.9 (10.9) | 56.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 312 | 474
  Male | 141 | 290 | 431
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 16 | 41 | 57
  Black or African American | 23 | 53 | 76
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 249 | 478 | 727
  Other | 13 | 26 | 39
  Mixed Race | 2 | 0 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 17 | 33 | 50
  Not Hispanic/Latino | 286 | 569 | 855
Background Therapy [Number; unit: participants]
  Diet Only | 38 | 74 | 112
  Diet + Atorvastatin 10 mg | 129 | 256 | 385
  Diet + Atorvastatin 80 mg | 73 | 146 | 219
  Diet + Atorvastatin 80 mg + Ezetimibe 10 mg | 63 | 126 | 189
Low-density Lipoprotein Cholesterol (LDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Cholesterol was measured by means of ultracentrifugation. Data are provided for the Full Analysis Set (all participants who were randomized and received at least 1 dose of study treatment).
  mg/dL | 104.0 (21.6) | 104.2 (22.1) | 104.1 (22.0)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the Full Analysis Set
  mg/dL | 179.1 (27.2) | 176.8 (27.5) | 177.6 (27.4)
Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the Full Analysis Set
  mg/dL | 125.6 (26.9) | 124.2 (25.6) | 124.6 (26.1)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the Full Analysis Set
  mg/dL | 87.5 (16.3) | 87.0 (16.3) | 87.2 (16.3)
Total Cholesterol/High Density Lipoprotein-Cholesterol (HDL-C) Ratio [Mean (Standard Deviation); unit: ratio] — Data are provided for the Full Analysis Set
  ratio | 3.603 (1.11) | 3.597 (1.04) | 3.599 (1.06)
Apolipoprotein B/Apolipoprotein A-1 Ratio [Mean (Standard Deviation); unit: ratio] — Data are provided for the Full Analysis Set
  ratio | 0.586 (0.170) | 0.593 (0.170) | 0.590 (1.70)
Lipoprotein(a) Concentration [Mean (Standard Deviation); unit: nmol/L] — Data are provided for the Full Analysis Set
  nmol/L | 89.3 (108.6) | 84.0 (98.5) | 85.8 (102.0)
Triglycerides Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the Full Analysis Set
  mg/dL | 127.8 (65.8) | 119.8 (63.2) | 122.5 (64.1)
High-density Lipoprotein Cholesterol (HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are providedfor the Full Analysis Set
  mg/dL | 53.5 (16.1) | 52.6 (15.5) | 52.9 (15.7)
Very Low-density Lipoprotein Cholesterol (VLDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Data are provided for the Full Analysis Set
  mg/dL | 21.5 (13.4) | 20.0 (11.4) | 20.5 (12.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C at Week 52
Description: Cholesterol was measured by means of ultracentrifugation.
Time Frame: Baseline and Week 52
Population: Full Analysis Set (all randomized subjects who received at least 1 dose of study drug).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
percent change | 6.83 (1.75) | -50.14 (1.24)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; The null hypothesis was that there was no mean difference in the percent change from Baseline at Week 52 in LDL-C between evolocumab 420 mg and placebo, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model; The model included treatment group, stratification factor, scheduled visit and the interaction of treatment with scheduled visit as covariates; LS Mean Treatment Difference = -56.97, 95% CI 2-sided [-61.08 to -52.85], Standard Error of Mean 2.10 — Treatment difference using placebo as the reference

2. Secondary Outcome: Change From Baseline in LDL-C at Week 52
Description: Cholesterol was measured by means of ultracentrifugation.
Time Frame: Baseline and Week 52
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
mg/dL | 5.1 (1.9) | -52.7 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model; The model includes treatment group, stratification factor, scheduled visit and the interaction of treatment with scheduled visit as covariates; LS Mean Treatment Difference = -57.8, 95% CI 2-sided [-62.3 to -53.3], Standard Error of Mean 2.3 — Treatment difference using placebo as the reference

3. Secondary Outcome: Percentage of Participants With an LDL-C Response at Week 52
Description: An LDL-C response is defined as LDL-C level < 70 mg/dL (1.8 mmol/L) at Week 52.
Time Frame: Week 52
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
percentage of participants | 6.4 [4.1 to 10.1] | 82.3 [78.8 to 85.3]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH test stratified by the stratification factor. For testing, non-achievement was imputed for participants with a missing value at Week 52; Treatment Difference = 75.8, 95% CI 2-sided [70.8 to 79.7] — Treatment difference using placebo as the reference

4. Secondary Outcome: Percent Change From Baseline in LDL-C at Week 12
Description: Cholesterol was measured by means of ultracentrifugation.
Time Frame: Baseline and Week 12
Population: Full Analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
percent change | 3.17 (1.31) | -54.35 (0.96)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; LS Mean Treatment Difference = -57.51, 95% CI 2-sided [-60.57 to -54.45], Standard Error of Mean 1.56 — Treatment difference using placebo as the reference

5. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 12
Time Frame: Baseline and Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
percent change | 2.85 (0.87) | -32.30 (0.63)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; LS Mean Treatment Difference = -35.15, 95% CI 2-sided [-37.19 to -33.11], Standard Error of Mean 1.04 — Treatment difference using placebo as the reference

6. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 52
Time Frame: Baseline and Week 52
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
percent change | 5.26 (1.16) | -28.18 (0.84)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; LS Mean Treatment Difference = -33.45, 95% CI 2-sided [-36.21 to -30.68], Standard Error of Mean 1.41 — Treatment difference using placebo as the reference

7. Secondary Outcome: Percent Change From Baseline in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) at Week 52
Time Frame: Baseline and Week 52
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
percent change | 8.44 (1.68) | -41.82 (1.21)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; LS Mean Treatment Difference = -50.27, 95% CI 2-sided [-54.25 to -46.28], Standard Error of Mean 2.03 — Treatment difference using placebo as the reference

8. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 52
Time Frame: Baseline and Week 52
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
percent change | 2.94 (1.41) | -41.26 (1.02)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; LS Mean Treatment Difference = -44.21, 95% CI 2-sided [-47.56 to -40.85], Standard Error of Mean 1.71 — Treatment difference using placebo as the reference

9. Secondary Outcome: Percent Change From Baseline in the Total Cholesterol/HDL-C Ratio at Week 52
Time Frame: Baseline and Week 52
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
percent change | 6.47 (1.37) | -30.67 (0.99)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; LS Mean Treatment Difference = -37.14, 95% CI 2-sided [-40.41 to -33.87], Standard Error of Mean 1.67 — Treatment difference using placebo as the reference

10. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A1 Ratio at Week 52
Time Frame: Baseline and Week 52
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
percent change | 4.46 (1.50) | -41.75 (1.09)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; LS Mean Treatment Difference = -46.21, 95% CI 2-sided [-49.79 to -42.63], Standard Error of Mean 1.82 — Treatment difference using placebo as the reference

11. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 52
Time Frame: Baseline and Week 52
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
percent change | -5.37 (1.62) | -27.72 (1.19)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; LS Mean Treatment Difference = -22.35, 95% CI 2-sided [-26.15 to -18.55], Standard Error of Mean 1.94 — Treatment difference using placebo as the reference

12. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 52
Time Frame: Baseline and Week 52
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
percent change | 8.99 (2.39) | -2.55 (1.72)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; LS Mean Treatment Difference = -11.54, 95% CI 2-sided [-17.21 to -5.86], Standard Error of Mean 2.89 — Treatment difference using placebo as the reference

13. Secondary Outcome: Percent Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C) at Week 52
Time Frame: Baseline and Week 52
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
percent change | 0.35 (0.90) | 5.77 (0.65)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; LS Mean Treatment Difference = 5.42, 95% CI 2-sided [3.28 to 7.56], Standard Error of Mean 1.09 — Treatment difference using placebo as the reference

14. Secondary Outcome: Percent Change From Baseline in Very Low-density Lipoprotein Cholesterol (VLDL-C) at Week 52
Description: Cholesterol was measured by means of ultracentrifugation.
Time Frame: Baseline and Week 52
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 302 | 599
percent change | 31.89 (4.69) | 2.74 (3.36)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; LS Mean Treatment Difference = -29.15, 95% CI 2-sided [-40.23 to -18.08], Standard Error of Mean 5.64 — Treatment difference using placebo as the reference

15. Secondary Outcome: Percent Change From Week 12 to Week 52 in LDL-C
Description: Cholesterol was measured by means of ultracentrifugation.
Time Frame: Week 12 and Week 52
Population: The Effect Durability Analysis Set included participants in the FAS who adhered to the scheduled study drug and had nonmissing LDL-C values at Baseline, Week 12 and Week 52.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 253 | 514
percent change | 2.57 (1.56) | 2.44 (1.14)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p = 0.94, ANCOVA; The ANCOVA model includes treatment group and stratification factor as covariates; LS Mean Treatment Difference = -0.14, 95% CI 2-sided [-3.76 to 3.48], Standard Error of Mean 1.84 — Treatment difference using placebo as the reference

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Evolocumab
Serious Adverse Events (participants affected / at risk) | 13/302 | 33/599
Other Adverse Events (participants affected / at risk) | 76/302 | 177/599
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=302) | Evolocumab (N=599)
Angina pectoris (Cardiac disorders) | 2 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 2
Exostosis of external ear canal (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Device breakage (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Biliary tract disorder (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Migraine with aura (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Breast prosthesis implantation (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=302) | Evolocumab (N=599)
Influenza (Infections and infestations) | 19 | 45
Nasopharyngitis (Infections and infestations) | 29 | 63
Upper respiratory tract infection (Infections and infestations) | 19 | 56
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.